CLINICAL TRIAL: NCT04304196
Title: Reducing Anxiety and Enhancing Quality of Life Among Caregivers of Prostate Cancer Survivors: Development and Evaluation of a Dyadic, Tailored, Web-based, Psychosocial and Physical Activity Self-management Programme
Brief Title: Tailored, wEb-based, Psychosocial and Physical Activity Self-Management PrOgramme
Acronym: TEMPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Mary's Research Center, Canada (Other)
Responsible Party: Principal Investigator, Sylvie Lambert, Principal Scientist, St. Mary's Research Center, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MP-CUSM-15-179
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Cancer of Prostate; Anxiety
Keywords: Caregiver; Self-directed online interventions; Coping; Self-management; Cancer; Physical activity
MeSH Terms: conditions — Prostatic Neoplasms; Anxiety Disorders; Neoplasms; Motor Activity | interventions — TEMPO

STUDY DESIGN:
Intervention Model Description: This pilot study is a multicenter, stratified, parallel, two-group randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEMPO (Experimental): These patients and caregivers will be able to access the TEMPO modules and will receive technical support to use it effectively. Patients will receive usual care throughout the study.
  Interventions: Other: TEMPO
- Control (Active Comparator): Patients will receive usual care throughout the study. Dyads in this group will not receive any information resources from the research team, but will have access to all of those available at their participating center (sites will be asked to provide a description of usual care practices). Participants will be given access to the TEMPO website after having completed their final questionnaire, as thanks for participating.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: TEMPO — TEMPO is designed as a 7- to 10-week, web-based intervention containing 5 modules to pace patient-caregiver dyads' learning, avoid information overload, and allow sufficient practice time in-between modules . Each module is organized along six key components: needs assessment, tailored information and skills training, goal setting and action planning, motivational and social support, monitoring, automated feedback, and addressing time demands. Overall, modules aim to a) increase dyads' confidence in using strategies to address key psychosocial issues in the acute survivorship phase (e.g., dealing with stress and worry, communicating with partner and family, uncertainty management) and b) assist dyads in developing the self-regulatory skills necessary to meet the physical activity guidelines. Each module specifies a series of online (i.e. didactic material and interactive worksheets) and offline activities (i.e. practicing the proposed skills).
  Other Names: Tailored, wEb-based, Psychosocial and Physical Activity Self-Management PrOgramme
  Arms: TEMPO
Other: Usual care — Patients will receive usual care throughout the study. Dyads in this group will not receive any information resources from the research team, but will have access to all of those available at their participating center (sites will be asked to provide a description of usual care practices). Participants will be given access to the TEMPO website after having completed their final questionnaire, as thanks for participating.
  Arms: Control

SUMMARY:
Caregivers of men with prostate cancer report high physical and emotional distress, and there is an urgent need to develop cost-effective programmes to prepare them for their roles. An online tool has been developed recently, aiming to offer a convenient, efficient, and potentially effective solution. However, pilot testing is required to evaluate this dyadic, Tailored, wEb-based, psychosocial and physical activity self-Management PrOgramme (called TEMPO) for caregivers of prostate cancer survivors. This study will assess TEMPO's acceptability, feasibility, cost, and potential efficacy, in addition to documenting the benefits (costs and outcomes) gained from involving both the caregiver and the patient in the intervention. A total of 80 patient-caregiver dyads will be recruited and randomized to a) TEMPO, or b) usual care. Acceptability, feasibility, and cost indicators will also be collected. Quality of life, anxiety, self-management skills, physical activity, self-efficacy, appraisal, and depression will also be assessed at baseline and 3 months post-baseline. In addition, intervention dyads will be invited to participate in an exit interview. This pilot study aims to assess the feasibility of the project, to inform the development and planning of a larger trial.

DETAILED DESCRIPTION:
BACKGROUND: Despite improvement in survival rates, a prostate cancer diagnosis still elicits negative reactions and confronts both patients and their partners and family caregivers (collectively referred to as 'caregivers') with a wide range of complex physical and psychosocial challenges. However, caregivers' support reduces the demands on the health care system and positively impacts on how well their loved ones adjust to the illness, their support comes at a particularly high cost to their own health and functioning. A recent review found that 16% to 68% of caregivers report needing more support to meet the challenges of their role. Such rates of unmet supportive care needs not only exceed those reported by the patients, but also further contribute to caregivers' burden and adversely impact on patients' quality of life (QOL). In light of caregivers' challenges, the first dyadic, Tailored, wEb-based, psychosocial and physical activity self-Management PrOgramme (called TEMPO) has been developed recently. TEMPO aims to increase patient-caregivers dyads' access to QOL-enhancing support and information, tailored to their needs. Due to the novel nature of this resource, no previous study has evaluated the usefulness of TEMPO.

OBJECTIVES: The goal of this pilot study is to inform the development and planning of a larger trial to evaluate the impact of TEMPO on key outcome measures for patients and caregivers. The primary objective of this pilot study is to (a) explore the feasibility and acceptability of the trial procedures and (b) estimate the cost-effectiveness of this intervention. The secondary objective is to estimate the clinical significance of using TEMPO on the primary and secondary outcomes.

METHODOLOGY: This pilot study is a multicenter, stratified, parallel, two-group RCT. Participating dyads will be randomized to receive (a) TEMPO with usual care or (b) usual care alone. Across participating sites, research assistants (RAs) will screen new patient records and confirm with clinicians whether the patients meet the medical eligibility. The clinician will then obtain interested patients' permission for a RA to approach them and provide further information, including a study brochure. If the potential participant(s) are interested, the RA will take them to a quiet/separate location to further explain the study, check eligibility using the eligibility checklist, and obtain consent. If it is not possible, at a minimum, the RA or hospital volunteer will get potential participants' contact information and their approval for a member of the research team to follow-up. Eligible and interested patients will complete an online consent form. If the caregiver is not present, the RA will provide study information to the patient and obtain his/her verbal consent to follow-up by phone within the next week to determine the caregiver's interest in the study. In addition, each site will display study posters giving potential participants the ability to self-refer.

A convenience sample of patients and their caregivers will be recruited from the , McGill University Health Centre (MUHC), Tom Baker Cancer Centre (TBCC), Vancouver General Hospital (VGH), and Sunnybrook Health Sciences Centre (SHSC).

Patient inclusion criteria are:

1. confirmed prostate cancer diagnosis (localized or advanced) within the past two years,
2. identified a primary caregiver willing to participate in the study,
3. is undergoing or has undergone active treatment (i.e., surgery, chemotherapy, radiotherapy, and/or hormonotherapy),
4. has access to the internet,
5. understands English or French. Eligible caregivers will be those identified by the patient as his primary source of support. Caregivers who were diagnosed with cancer in the previous year, or who are currently receiving treatment for cancer will be excluded. Patients and caregivers also need to be able to understand English or French.

SIGNIFICANCE: The ability of caregivers to maintain their QOL despite the stressors they face is undermined by limited access to the support needed. This study will evaluate the first dyadic, tailored, web-based, psychosocial and physical activity self-management programme, and address a significant research gap by documenting its acceptability, feasibility. In addition, this study will estimate its potential clinical significance.

ELIGIBILITY:
Inclusion Criteria (patient):

* confirmed prostate cancer diagnosis (localized or advanced) within the past two years,
* identified a primary caregiver willing to participate in the study,
* is undergoing or has undergone active treatment (i.e., surgery, chemotherapy, radiotherapy, and/or hormonotherapy),
* has access to the internet,
* understands English

Exclusion Criteria (patient):

* medical contraindications to participate in moderate physical activity

Inclusion Criteria (caregiver):

* identified as a primary caregiver by an eligible patient willing to participate in the study
* understands English

Exclusion Criteria (caregiver):

* diagnosed with cancer in the previous year
* currently receiving treatment for cancer will be excluded
* medical contraindications to participate in moderate physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-05-29 (Actual); Study Completion 2021-05-29 (Actual)

PRIMARY OUTCOMES:
Consent and follow-up rates | From recruitment launch to completion of follow-up (12 months)
  Number of consenting dyads per week over the recruitment period
Data completion rate | At T2: 13 weeks
  Investigators will report on rates of missing data from pilot baseline and follow-up questionnaires.
Fidelity of intervention completion | At T2: 13 weeks
  Logs will be used to evaluate completion of intervention, as per protocol (e.g., number of log-ins, time spent, modules completed).
Rate of tool use | At T2: 13 weeks
  A 26-item questionnaire was developed by the team to evaluate the tool use. Each statement is scored using a 7-point likert scale, ranging from "completely disagree" to "completely agree". The total score is calculated by combining each individual item score. The total score ranges from 0 to 156. Higher score means better outcomes.
Service Usability Scale | At T2: 13 weeks
  The Service Usability Scale will be used. The score (1-5 Likert Scale, ranging from "strongly disagree" to "strongly agree") of the 10 statements will be combined into a final note (between 10 and 50). Higher score means better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Lambert, PhD, Principal Investigator — McGill University
Locations (1):
- St Mary's Hospital Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lambert SD, Duncan LR, Ellis J, Robinson JW, Sears C, Culos-Reed N, Matthew A, De Raad M, Schaffler JL, Mina DS, Saha-Chaudhuri P, McTaggart-Cowan H, Peacock S. A study protocol for a multicenter randomized pilot trial of a dyadic, tailored, web-based, psychosocial, and physical activity self-management program (TEMPO) for men with prostate cancer and their caregivers. Pilot Feasibility Stud. 2021 Mar 20;7(1):78. doi: 10.1186/s40814-021-00791-6. PMID 33743804